CLINICAL TRIAL: NCT02146703
Title: Phase II Trial of Gemcitabine and S-1 for Patients With Advanced Biliary Tract Cancer
Brief Title: Gemcitabine and S-1 for Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-0501
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Biliary Tract Neoplasm
Keywords: biliary tract neoplasm; gemcitabine; S-1
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine and S-1 (Experimental)
  Interventions: Drug: Gemcitabine, and S-1

INTERVENTIONS:
Drug: Gemcitabine, and S-1 — Treatment will be delivered as a 3-week cycle.
  1. Gemcitabine 1000 mg/m2 iv on day 1, 8
  2. S-1 60 mg/day po on day 1-14
  Other Names: Gemzar; TS-1

SUMMARY:
This study will conduct a phase II study of gemcitabine and S-1 as first-line chemotherapy in patient with advanced biliary tract cancer

DETAILED DESCRIPTION:
Biliary-tract cancer (BTC) is invasive carcinoma that originates from the epithelial lining of the gallbladder and bile ducts. BTC include cholangiocarcinoma (intrahepatic, perihilar, and distal biliary-tree tumor) and carcinoma arising from the gallbladder.

Surgical resection of the primary tumor is potentially curative for BTC, but less than a quarter of patients are eligible for resection at presentation. Systemic chemotherapy is the principal treatment method for patients with unresectable or metastatic BTC.

Gemcitabine is a promising agent, which has shown efficacy in biliary tract cancer. As a single-agent therapy, gemcitabine shows response rates of 8-36% in BTC[4]. In phase II trials with patients in advanced BTC, gemcitabine in combination with capecitabine or platinum analogues produced objective response rates of 26-50%.

The ABC-02 study reported a significant survival advantage for gemcitabine and cisplatin over gemcitabine alone in patients with advanced BTC (median overall survival 11.7 vs. 8.1 months; P < 0.001).

Oral anticancer drug S-1 consists of the 5-FU prodrug tegafur with two biochemical modulators, 5-chloro-2,4-dihydroxypyridine (CDHP) and potassium oxonate (Oxo). S-1 monotherapy is active against advanced BTC with objective response rates of 21-35%, and phase II trials of S-1 in combination with gemcitabine reported objective response rates of 20-36%. Differences between trials in the doses and administration schedules of gemcitabine and S-1 may be reflected in the ranges of efficacy, dose-intensity, and rates of toxicity observed.

Even though the efficacy of gemcitabine and S-1 combination is evident for patients with advanced BTC in previous phase II trials, there was no clinical study investigating the efficacy of gemcitabine and S-1 combination for patients with advanced BTC when this study was started. Therefore, we conducted a phase II study to evaluate gemcitabine and S-1 combination as first-line chemotherapy for patients with advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced, metastatic adenocarcinoma arising from the intra- and extrahepatic biliary ducts or gallbladder
* Initially diagnosed or recurred
* At least one bidimensionally measurable lesion, defined as at least 1x1cm with clearly defined margins on physical examination, on 3-dimentional CT, MRI, or PET-CT
* Age ≥18 and ≤70 years
* Estimated life expectancy ≥3 months
* ECOG performance status ≤2
* Adequate bone marrow function (WBCs ≥4,000/µL or absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL),
* Adequate kidney function (creatinine ≤1.4 mg/dL)
* Adequate liver function (bilirubin ≤1.8 mg/dL, transaminase levels ≤100mg/dL)
* Written informed consent

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Previous history of chemotherapy (exception : adjuvant chemotherapy)
* Presence of CNS metastasis, psychosis, or seizure
* Obvious bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Past or concurrent history of neoplasm other than biliary adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-08; Primary Completion 2010-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate | 1 year

SECONDARY OUTCOMES:
Progression free survival, median overall survival, disease control rate, and over grade 3 hematologic toxicities (neutropenia, thrombocytopenia, and febrile neutropenia) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Medical Center, Anyang, South Korea

REFERENCES:
- [Background] Oertli D, Herzog U, Tondelli P. Primary carcinoma of the gallbladder: operative experience during a 16 year period. Eur J Surg. 1993 Aug;159(8):415-20. PMID 8218552
- [Background] de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999 Oct 28;341(18):1368-78. doi: 10.1056/NEJM199910283411807. No abstract available. PMID 10536130
- [Background] Thongprasert S. The role of chemotherapy in cholangiocarcinoma. Ann Oncol. 2005;16 Suppl 2:ii93-6. doi: 10.1093/annonc/mdi712. No abstract available. PMID 15958484
- [Background] Hezel AF, Zhu AX. Systemic therapy for biliary tract cancers. Oncologist. 2008 Apr;13(4):415-23. doi: 10.1634/theoncologist.2007-0252. PMID 18448556
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Shirasaka T, Shimamato Y, Ohshimo H, Yamaguchi M, Kato T, Yonekura K, Fukushima M. Development of a novel form of an oral 5-fluorouracil derivative (S-1) directed to the potentiation of the tumor selective cytotoxicity of 5-fluorouracil by two biochemical modulators. Anticancer Drugs. 1996 Jul;7(5):548-57. doi: 10.1097/00001813-199607000-00010. PMID 8862723
- [Background] Ueno H, Okusaka T, Ikeda M, Takezako Y, Morizane C. Phase II study of S-1 in patients with advanced biliary tract cancer. Br J Cancer. 2004 Nov 15;91(10):1769-74. doi: 10.1038/sj.bjc.6602208. PMID 15505626
- [Background] Furuse J, Okusaka T, Boku N, Ohkawa S, Sawaki A, Masumoto T, Funakoshi A. S-1 monotherapy as first-line treatment in patients with advanced biliary tract cancer: a multicenter phase II study. Cancer Chemother Pharmacol. 2008 Oct;62(5):849-55. doi: 10.1007/s00280-007-0673-7. Epub 2008 Jan 23. PMID 18214482
- [Background] Sasaki T, Isayama H, Nakai Y, Ito Y, Kogure H, Togawa O, Toda N, Yasuda I, Hasebe O, Maetani I, Sasahira N, Hirano K, Tsujino T, Tada M, Omata M. Multicenter, phase II study of gemcitabine and S-1 combination chemotherapy in patients with advanced biliary tract cancer. Cancer Chemother Pharmacol. 2010 May;65(6):1101-7. doi: 10.1007/s00280-009-1115-5. Epub 2009 Aug 26. PMID 19707761
- [Background] Kanai M, Yoshimura K, Tsumura T, Asada M, Suzuki C, Niimi M, Matsumoto S, Nishimura T, Nitta T, Yasuchika K, Taura K, Mori Y, Hamada A, Inoue N, Tada S, Yanagihara K, Yazumi S, Osaki Y, Chiba T, Ikai I, Fukushima M, Uemoto S, Hatano E. A multi-institution phase II study of gemcitabine/S-1 combination chemotherapy for patients with advanced biliary tract cancer. Cancer Chemother Pharmacol. 2011 Jun;67(6):1429-34. doi: 10.1007/s00280-010-1443-5. Epub 2010 Sep 2. PMID 20811895
- [Background] Sasaki T, Isayama H, Nakai Y, Ito Y, Yasuda I, Toda N, Kogure H, Hanada K, Maguchi H, Sasahira N, Kamada H, Mukai T, Okabe Y, Hasebe O, Maetani I, Koike K. A randomized phase II study of gemcitabine and S-1 combination therapy versus gemcitabine monotherapy for advanced biliary tract cancer. Cancer Chemother Pharmacol. 2013 Apr;71(4):973-9. doi: 10.1007/s00280-013-2090-4. Epub 2013 Jan 26. PMID 23355041
- [Background] Morizane C, Okusaka T, Mizusawa J, Takashima A, Ueno M, Ikeda M, Hamamoto Y, Ishii H, Boku N, Furuse J. Randomized phase II study of gemcitabine plus S-1 versus S-1 in advanced biliary tract cancer: a Japan Clinical Oncology Group trial (JCOG 0805). Cancer Sci. 2013 Sep;104(9):1211-6. doi: 10.1111/cas.12218. Epub 2013 Jul 25. PMID 23763511